CLINICAL TRIAL: NCT00765687
Title: A Multi-center Observational Clinical Study of Screening of Non-small-cell Lung Cancer With Bone Metastasis and Efficacy and Safety of Those Receiving Bisphosphonates
Brief Title: Screening Non Small Cell Lung Cancer With Bone Metastasis and Efficacy and Safety Research of Receiving Bisphosphonates
Acronym: BLEST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Li Zhang, Profressor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CZOL446ECN07
Record Dates: First submitted 2008-09-29; First posted 2008-10-03 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2011-12

CONDITIONS: Non-small Cell Lung Cancer; Bone Metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Observation (No Intervention)
  Interventions: Drug: bisphosphates

INTERVENTIONS:
Drug: bisphosphates — any bisphosphate, repeated every 4 weeks for up to 24 months. Co-administration with Zometa: Calcium 500 mg + vitamin D 400-500 IU daily

SUMMARY:
A multicenter Prospective Study to assess the screening methods, parameter of NTX and the efficacy and safety of zoledronic acid treatment in addition to anti-tumor therapy in patients of non-small cell cancer with bone metastasis in china.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18, either sex
2. Histologically confirmed non-small cell cancer
3. One bone metastasis at least confirmed by image(X ray,CT or others)
4. Without receiving zoledronic acid
5. Life expectancy > 6 M
6. ECOG <= 2
7. Signed ICF

Exclusion Criteria:

1. Women who are pregnant or in lactation
2. Patients with hyperostosis
3. with brain metastasis(exception of those without symptom or with Metastasis Lesions under controlled
4. Previous or current treatment with any other bisphosphonates, bone- protecting, cytotoxic or targeted therapy
5. Severe co-morbidity of any type that may interfere with assessment of the patient for the study -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2008-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Skeleton-related event | 24 months

SECONDARY OUTCOMES:
overall survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Li, Master, Principal Investigator — Cancer Center of Sun Yat-Sen University (CCSU)
Locations (1):
- SunYat-senU, Guangzhou, Guangdong, China